CLINICAL TRIAL: NCT03860376
Title: Personalized Ex Vivo Drug Screening and Genomics Profiling to Guide Individualized Treatments for Children With Relapsed or Refractory Solid Tumors and Leukemias
Brief Title: Ex Vivo Drug Sensitivity Testing and Mutation Profiling
Status: Completed | Type: Observational
Sponsor: Florida International University (Other)
Collaborators: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Principal Investigator, Diana Azzam, PhD, Assistant Professor, Florida International University
Other Study IDs: 1186919; 8LA05 (Other Grant/Funding Number: Florida Department of Health-Live Like Bella Foundation)
Record Dates: First submitted 2019-02-11; First posted 2019-03-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Large Cell Lymphoma; Refractory Childhood Acute Lymphoblastic Leukemia; Refractory Childhood Hodgkin Lymphoma; Refractory Childhood Malignant Germ Cell Neoplasm; Recurrent Childhood Brain Tumor; Recurrent Childhood Brainstem Glioma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Ependymoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Gliosarcoma; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive
Keywords: ex vivo drug sensitivity assay; genomic profiling
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Familial ependymoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Perform molecular and functional drug testing on blood, biopsy, bone marrow and tumor samples at relapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chemorefractory or relapsed patients: We intend to enroll chemorefractory or relapsed pediatric patients with all types of cancers where tumor tissue would be available for ex vivo drug screening and genomic profiling. The results of the drug sensitivity assay and genetic screening will be used to inform treating physician about patient-specific drug sensitivity or resistance guiding best therapy choices.

SUMMARY:
This study is a prospective, non-randomized feasibility study. Freshly isolated tumor cells from patients will be screened using state-of-the-art viability assay designed for ex vivo high-throughput drug sensitivity testing (DST). In addition, genetic information will be obtained from cancer and normal (germline) tissue and correlated with drug response. This study will provide the platform for informing treating physician about individualized treatment options. The main outcome of this study will be the proportions of the patients whose treatment was guided by the personalized medicine approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: The primary objective of the study is to determine feasibility of providing pediatric cancer patients with access to personalized treatment options and clinical management recommendations based on ex vivo drug sensitivity testing (DST) and genomic profiling.

SECONDARY OBJECTIVE: The secondary objective of the study is to compare individual outcomes (response and disease-free survival) in patients with pediatric cancers treated with DST-guided therapy as compared to non-DST guided (conventional) therapy.

EXPLORATORY OBJECTIVE: To explore associations between genetic abnormalities in malignancies and ex vivo drug response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or younger at the time of enrollment on this study of any gender, race or ethnicity.

  * Subjects with suspected or confirmed diagnosis of recurrent or refractory cancer
  * Subjects who are scheduled for or have recently had biopsy or tumor excised (solid tumors) or bone marrow aspirate (blood cancers)
  * Subjects willing to have a blood draw or buccal swab done for the purposes of genetic testing
  * Subjects or their parents or legal guardians willing to sign informed consent
  * Subjects aged 7 to 17 willing to sign assent

Exclusion Criteria:

* Subjects who do not have malignant tissue available and accessible
* The amount of excised malignant tissue is not sufficient for the ex vivo drug testing and/or genetic profiling.
* Patients with newly diagnosed tumors and tumors that have high (>90%) cure rate with safe standard therapy.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chemorefractory and/or relapsed pediatric cancer patients with no alternative treatment options.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that receive DST-guided treatmens | Up to 4 years
  This study will be considered successful (feasibility demonstrated) if it is possible to choose and initiate a monotherapy or combination drug regimen based on functional and/or genomics data within 4 weeks in at least 16 out of 25 patients (64%).
  To achieve at least 90% power, the null hypothesis will be rejected when at least 16 out of 25 patients receive treatment recommendations through functional and/or genomics data within 4 weeks on the study.
  With that outcome, we would have 95% confidence that the true feasibility rate is at least 30% (95% CI: 0.425, 1).

SECONDARY OUTCOMES:
Assessing Objective Response Rate | Up to 4 years
  We will assess changes in cohort Objective Response Rate (ORR) by comparing ORR in patients treated with FPM-guided therapy versus ORR in patients treated with non-FPM guided conventional therapy (standard of care)
Assessing Progression-Free Survival (PFS) | Up to 4 years
  We will assess changes in cohort PFS by comparing PFS in patients treated with FPM-guided therapy versus PFS in patients treated with non-FPM guided conventional therapy (standard of care)
Assessing Previous vs Trial PFS Ratio (PFS2/PFS1) | Up to 4 years
  We will assess changes in PFS from each patient's previous treatment versus their PFS from the treatment assigned during the trial. Assessments will be made both in the FPM-guided cohort and the non-FPM-guided conventional therapy cohort. Analysis will include both the raw ratio as well as the number of incidences of 30% improved PFS on trial versus previous regimen (PFS2/PFS1 > 1.3x).

CONTACTS AND LOCATIONS:
Overall Officials: Diana Azzam, PhD, Principal Investigator — Florida International University; Daria Salyakina, PhD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States

REFERENCES:
- [Result] Acanda De La Rocha AM, Fader M, Coats ER, Espinal PS, Berrios V, Saghira C, Sotto I, Shakya R, Janvier M, Khatib Z, Abdella H, Bittle M, Andrade-Feraud CM, Guilarte TR, McCafferty-Fernandez J, Salyakina D, Azzam DJ. Clinical Utility of Functional Precision Medicine in the Management of Recurrent/Relapsed Childhood Rhabdomyosarcoma. JCO Precis Oncol. 2021 Oct 27;5:PO.20.00438. doi: 10.1200/PO.20.00438. eCollection 2021. No abstract available. PMID 34738048
- [Derived] Acanda De La Rocha AM, Berlow NE, Fader M, Coats ER, Saghira C, Espinal PS, Galano J, Khatib Z, Abdella H, Maher OM, Vorontsova Y, Andrade-Feraud CM, Daccache A, Jacome A, Reis V, Holcomb B, Ghurani Y, Rimblas L, Guilarte TR, Hu N, Salyakina D, Azzam DJ. Feasibility of functional precision medicine for guiding treatment of relapsed or refractory pediatric cancers. Nat Med. 2024 Apr;30(4):990-1000. doi: 10.1038/s41591-024-02848-4. Epub 2024 Apr 11. PMID 38605166